CLINICAL TRIAL: NCT06355323
Title: Bronchiectasis Prevalence in Patients With Primary Humoral Immunodefiency in Champagne-Ardenne Region, France
Acronym: PREDDICHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PT22020
Record Dates: First submitted 2023-02-24; First posted 2024-04-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Immunodeficiency; Common Variable Immunodeficiency; Igg Subclass Deficiency; Selective IgM Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; IgG Deficiency | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: Blood test; Other: chest CT scan

INTERVENTIONS:
Other: Blood test — Blood test
Other: chest CT scan — chest CT scan

SUMMARY:
Primary humoral immunodeficiency (PHID), such as common variable immunodefiency, are the most common symptomatic primary immunodeficiency in adults, in France. Patients are more prone to infections (particularly bacterial upper and lower respiratory tract infections), auto-immunity and atopic manifestations. Morbidity and mortality in PHID are mainly linked to the presence of bronchiectasis, which can lead to infections and to chronic respiratory failure. However, bronchiectasis in these patients can be asymptomatic for a long time. There is no known predictive factors to identify patients more susceptible to develop bronchiectasis and notably, there was no link between the number of previous infectious episodes and bronchiectasis. A marked IgM deficiency and switched memory B cell deficiency might be associated with bronchiectasis.

Thoracic CT-scan is recommended at PHID diagnosis but there is no guideline for follow-up, thus leading to bronchiectasis being under-diagnosis or leading to delayed diagnosis

DETAILED DESCRIPTION:
Common variable immunodeficiency (CVID) and other antibody deficiencies like immunoglobin G subclass deficiency and selective IgM deficiency are the most frequent clinically significant primary immunodeficiencies (PID) in adults. Prevalence in France in 2009 was 2.11/100.000 people.

These immunodeficiencies are characterized by a significant decrease in serum immunoglobulin concentrations and antibodies production. In some patients, qualitative and/or quantitative alterations in B cells repertoire and sometimes in T cells repertoire are observed. Consequently, patients are more prone to bacterial infections, respiratory manifestations, auto-immune diseases, atopic manifestations, neoplastic complications. Respiratory manifestations are the main complication responsible for the morbidity and mortality in PHID. Bronchiectasis are one of the observed pulmonary complications. It is characterized by pathological and permanent dilatation of the airways, as demonstrated by a thoracic CT-scan. Its frequency varies from a study to another, ranging from 20% to 60% in different PHID populations. Some patients with bronchiectasis can be asymptomatic, while others can present daily symptoms of cough and sputum production with periodic worsening of their symptoms (exacerbations). It can lead to chronic respiratory failure, more infectious complications and altered quality of life. Moreover, mortality in patients with bronchiectasis (whatever the cause) is twice as high than in general population.

A thoracic CT-scan is therefore recommended at PHID diagnosis. However, there is no recommendation concerning screening of this complication during follow-up.

Pathophysiology of bronchiectasis in general is described as a cycle of events promoting impaired mucociliary clearance and retention of airways secretions, leading to chronic infection and thus to inflammatory response, leading to abnormal remodeling oh the airways.

To date, it is not known if some PHID patients are more prone to developing bronchiectasis. There is no statistical link with the number of past infectious events. Some studies suggested that patients with lower IgM concentration or lower switched memory B cell might be more at risk.

Concerning T-cell subset, polarization of CD4 T helper cells response as well as T follicular helper implication might be of interest. Indeed, in auto-immune manifestations in patients with primary immunodeficiency, T follicular helper cells (T cells implied in regulation of B -cells response in germinal centers) are sometimes impaired.

Another interesting phenomenon has been described in chronic obstructive pulmonary disease (another pulmonary disease, presenting similar clinical and pathophysiological mechanisms with bronchiectasis), where lung-infiltrating inflammatory cells secrete proteases participating in elastin breakdown a specific marker of elastin degradation genesis of elastin-derived peptides. These peptides modulate CD4+ T cell (T helper) response and pro-inflammatory cytokine production. As inflammatory response in patients with PHID can differ from immunocompetent patients, modulation of pro-inflammatory T helper cell response by elastin-derived peptides might also be different, participating in the abnormal remodeling of the airways.

In the Champagne-Ardenne region, PHID prevalence is high (5.37/100.000 habitants), however, we do not have data concerning bronchiectasis prevalence in this population and its repercussion on respiratory function and quality of life for our patients. Moreover, a better understanding of pathophysiology and factors associated with the presence of bronchiectasis may lead to better and more personalized care (diagnostic and therapeutic).

ELIGIBILITY:
inclusion criteria :

* Patients with primary humoral immunodeficiency defined as following :

  * Common variable immunodeficiency : Marked decreased in IgG seric concentration < 5 g/L and in IgA seric concentration or IgM seric concentration (-2SD), without secondary cause
  * IgG subclass deficiency : marked decrease (-2SD) in at least one IgG subclass (IgG1, 2, 3 et 4) with or without IgA or IgM deficiency
  * Selective IgM Deficiency : isolated decrease un IgM seric concentration <0.3g/L, without IgG or IgA deficiency
* Adult patients
* Patients with or without previously identified pulmonary complications
* Patients agreeing to participate to the study
* Patients insured under the French social security system

Non-inclusion criteria :

* Patients< 18 years of age
* Patients protected by law
* Patients for whom CT scan is not feasible (claustrophobia, obesity…)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Thoracic CTscan | Day 0
  non-contrast thin-section thoracic CT-scan, after negative urine pregnancy test for women of childbearing age, allowing to detect presence of bronchiectasis and if present the severity index (Bhalla score)

SECONDARY OUTCOMES:
Pulmonary Function Test | Day 0
  Measures with plethysmography : Forced Expiratory volume
Pulmonary Function Test | Day 0
  Measures with plethysmography : DLCO
Pulmonary Function Test | Day 0
  Measures with plethysmography : Total Lung Capacity
Pulmonary Function Test | Day 0
  Measures with plethysmography : Residual Volume
Pulmonary Function Test | Day 0
  Measures with plethysmography : Functional Residual Capacity
Pulmonary Function Test | Day 0
  Measures with plethysmography : Vital Capacity
6 minutes walking test | Day 0
  measurement of maximal distance walked in 6 minutes
6 minutes walking test | Day 0
  saturation in oxygen (SpO2)
6 minutes walking test | Day 0
  Borg index after test
6 minutes walking test | Day 0
  Borg index before test
Quality of life questionnaires | Day 0
  SF-36
Quality of life questionnaires | Day 0
  BHQ
Immunophenotyping | Day 0
  description of some circulating B and T cells subsets
Biochemical factors : desmosine seric concentration | Day 0
  Measurement of desmosine seric concentration (a specific marker of elastin degradation)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France